CLINICAL TRIAL: NCT06661408
Title: The Effects of Video-Based and Practical Newborn Bathing Education Provided to Primiparous Pregnant Women During the Third Trimester on Knowledge, Anxiety, and Bonding During the First Bath: a Randomized Controlled Trial
Acronym: NewbornBathing
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Çağla KILIÇ, Research Assistant, Kahramanmaras Sutcu Imam University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 185; TUBITAK or KSU BAP (Other: TUBITAK or KSU BAP)
Record Dates: First submitted 2024-09-17; First posted 2024-10-28 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-08

CONDITIONS: Newborn Bathing; Primiparous Pregnant Women; Anxiety; Bonding; Knowledge
Keywords: Newborn; Bathing; Primipar; Education
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Randomized controlled experimental research
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control Group (No Intervention): Pregnant women in the control group will be subjected to the routine hospital protocol without any other intervention. Pregnant women in this group are verbally informed about bathing during outpatient clinic follow-ups. After completing the post-test questions, the newborn bath application video will be transmitted to the women in this group on their phones and the disadvantageous situation of this group will be tried to be reduced.
- Intervention group 1 (Experimental): The women assigned to this group will be shown the newborn bath application video prepared by the researchers in groups of 2-4 people in the form of a projection presentation.
  Interventions: Behavioral: Intervention group 1
- Intervention group 2 (Experimental): In groups of 2, the researcher will first explain the stages of newborn bathing application by the researcher in the form of a projection presentation, and then the pregnant women will be provided to perform the newborn bathing application on the newborn bathing model and tools simultaneously with the researcher.
  Interventions: Behavioral: Intervention group 2

INTERVENTIONS:
Behavioral: Intervention group 1 — The women assigned to this group will be shown the newborn bath application video prepared by the researchers in groups of 2-4 people in the form of a projection presentation.
  Arms: Intervention group 1
Behavioral: Intervention group 2 — In groups of 2, the researcher will first explain the stages of newborn bathing application by the researcher in the form of a projection presentation, and then the pregnant women will be provided to perform the newborn bathing application on the newborn bathing model and tools simultaneously with the researcher.
  Arms: Intervention group 2

SUMMARY:
This study will be conducted in a randomized controlled experimental research design with pretest, posttest control group.

DETAILED DESCRIPTION:
This study will be conducted in a randomized controlled experimental research design with pretest, posttest control group.

ELIGIBILITY:
Inclusion Criteria:

* Can speak and understand Turkish,
* 18 years of age or older,
* Literate,
* Primiparous,
* In the third trimester of pregnancy,
* A singleton pregnancy,
* No psychiatric illness,
* Who have not received any training on newborn bathing before,
* Her baby was not diagnosed with a fetal anomaly,
* With a smartphone and internet,
* Residing in the province of Kahramanmaras and
* Who agreed to participate in the research

Exclusion Criteria:

* Preterm labor (<37 weeks gestation),
* Stillbirth,
* The baby needs intensive care or is hospitalized,
* The baby has a low birth weight (<2500 grams),
* The one whose baby's first bath was given by someone else,
* A newborn bathing program was organized at the pregnancy school.
* Wishing to leave at any stage of the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2024-12-15 (Estimated); Primary Completion 2025-07-15 (Estimated); Study Completion 2025-08-15 (Estimated)

PRIMARY OUTCOMES:
Knowledge Level of Mothers on Newborn Bathing | average 3 months
  The Newborn Bathing Knowledge Test was developed by the researchers based on the literature to determine the knowledge levels of mothers about newborn bathing. In the knowledge test, there are a total of 20 questions under 10 main topics including "bath time, bathing materials, ambient temperature, water temperature, umbilical cord care, soap and shampoo use, maintaining newborn body temperature, bathing procedure sequence, safety during bathing, drying after bathing and dressing". The questions were prepared in multiple-choice and true/false design, and each question had only one correct answer. The women's answers to the questions were evaluated after the completion of the test and each correctly answered question was evaluated as five points and the total score ranged from 0-100. The higher the score obtained from the knowledge test, the higher the women's level of knowledge about newborn bathing.
Anxiety level of women | average 3 months
  Anxiety level of women will be assessed by using Spielberger's State Anxiety Inventory. The scale was developed to measure the state anxiety levels of normal and abnormal individuals and adapted into Turkish by Öner and Le Compte. It is a self-assessment type scale consisting of short statements. The State Anxiety Inventory was developed to measure a person's anxiety at a specific moment and consists of 20 items. In the evaluation of the scale, it is accepted that those who score below 36 have no anxiety, those who score between 37 and 42 have mild anxiety and those who score 42 and above have high anxiety.
Womens bonding levels | average 3 months
  Womens bonding level will be assessed using the Postpartum Bonding Questionnaire (PBQ). The PBQ was first developed to assess mother-infant attachment. It was revised to identify problems in the mother-infant relationship. The scale was adapted into Turkish by Dişsiz et al. in 2024. The six-point Likert-type scale has 21 items to measure the mothers attachment to the infant within a year. As the score obtained from the scale increases, the mothers bonding to the baby decreases.

CONTACTS AND LOCATIONS:
Locations (1):
- Kahramanmaras Sutcu Imam University, Kahramanmaraş, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] WHO Recommendations on Postnatal Care of the Mother and Newborn. Geneva: World Health Organization; 2013 Oct. Available from http://www.ncbi.nlm.nih.gov/books/NBK190086/ PMID 24624481
- [Background] Sarkar R, Basu S, Agrawal RK, Gupta P. Skin care for the newborn. Indian Pediatr. 2010 Jul;47(7):593-8. doi: 10.1007/s13312-010-0132-0. PMID 20683112
- [Background] Roxanne B, Laura VDB, Yannic VG, Natacha VC, Luka VL, Kuipers YJ. Validation of the postpartum bonding questionnaire: A cross-sectional study among Flemish mothers. Midwifery. 2022 Apr;107:103280. doi: 10.1016/j.midw.2022.103280. Epub 2022 Feb 8. PMID 35182820
- [Background] Öner N, Le Compte A. Süreksiz Durumluk/Sürekli Kaygı Envanteri El Kitabı. s: 1-26, 1. Basım Boğaziçi Üniversitesi Yayınları, İstanbul, 1983.
- [Background] Keten Edis E. Sağlık & Bilim 2022: Hemşirelik- IV. s. 95-103, 1. Basım, Efe Akademik Yayıncılık, İstanbul, 2022.
- [Background] Kayom VO, Kakuru A, Kiguli S. Newborn Care Practices among Mother-Infant Dyads in Urban Uganda. Int J Pediatr. 2015;2015:815938. doi: 10.1155/2015/815938. Epub 2015 Dec 2. PMID 26713096
- [Background] Getachew G, Ibrahim IM, Mulugeta Y, Ahmed KY. Early newborn bathing and associated factors among mothers in Afar Region, Northeast Ethiopia. J Trop Pediatr. 2022 Dec 5;69(1):fmac117. doi: 10.1093/tropej/fmac117. PMID 36625889
- [Background] Garcia Bartels N, Mleczko A, Schink T, Proquitte H, Wauer RR, Blume-Peytavi U. Influence of bathing or washing on skin barrier function in newborns during the first four weeks of life. Skin Pharmacol Physiol. 2009;22(5):248-57. doi: 10.1159/000235552. Epub 2009 Aug 18. PMID 19690450
- [Background] Dissiz M, Bayri Bingol F, Demirgoz Bal M, Karacam Yilmaz ZD, Karakoc A, Bilgin Z. The Turkish version of the Postpartum Bonding Questionnaire (PBQ): Examination of the validity and reliability and scale structure. J Pediatr Nurs. 2024 Jul-Aug;77:131-139. doi: 10.1016/j.pedn.2024.03.012. Epub 2024 Mar 21. PMID 38518689
- [Background] Dağoğlu T, Ovalı F. Yenidoğanın cilt bakımı. Neonatoloji. s.167-74, 2. Basım, Nobel Tıp Kitabevleri, İstanbul, 2007.
- [Background] Çalışır H, Güler F. Riskli Yenidoğanların cilt bakımında kanıta dayalı uygulamalar. Türkiye Klinikleri Hemşirelik Bilimleri Dergisi 2011; 3(2).
- [Background] Brockington IF, Oates J, George S, Turner D., Vostanis P, Sullivan M, ve ark. Screening questionnaire for mother-infant bonding disorders. Archives Of Women's Mental Health 2001; 3(4):133-140.
- [Background] Brandon D, Hill CM, Heimall L, Lund CH, Kuller J, McEwan T, New K. Neonatal skin care: evidence-based clinical practice guideline. Washington DC: Association of Women's Health, Obstetric and Neonatal Nurses 2018.
- [Background] Boran S, Kahriman İ, Polat SD. Exploring newborn bathing practices among mothers in the postpartum period. Genel Sağlık Bilimleri Dergisi 2024; 6(2):239-254.
- [Background] Blume-Peytavi U, Cork MJ, Faergemann J, Szczapa J, Vanaclocha F, Gelmetti C. Bathing and cleansing in newborns from day 1 to first year of life: recommendations from a European round table meeting. J Eur Acad Dermatol Venereol. 2009 Jul;23(7):751-9. doi: 10.1111/j.1468-3083.2009.03140.x. PMID 19646134
- [Background] American Academy of Pediatricks 2023. https://www.healthychildren.org/English/ages-stages/baby/bathing-skin-care/Pages/Bathing-Your-Newborn.aspx: Erişim Tarihi: 19.08.2024.